CLINICAL TRIAL: NCT05157334
Title: Can Manipulation of the Vagus Nerve Through Deep Breathing and Transcutaneus Electrical Nerve Stimulation Modulate Heart Rate Variability?
Brief Title: The Effect of Deep Breathing and Transcutaneus Electrical Nerve Stimulation on Heart Rate Variability
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Aalborg University Hospital (Other)
Collaborators: Aalborg University (Other)
Responsible Party: Principal Investigator, Salome Kristensen, Clinical associate professor, Priniciple investigator, MD, PhD, Aalborg University Hospital
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Basic Science
Other Study IDs: N-20210002
Record Dates: First submitted 2021-11-02; First posted 2021-12-15 (Actual); Last update posted 2021-12-15 (Actual); Status verified 2021-12

CONDITIONS: Rheumatoid Arthritis; Systemic Lupus Erythematosus; Healthy Participants
Keywords: Heart rate variability; Deep breathing; Transcutaneous vagus nerve stimulation; Vagus nerve stimulation; Breathing exercises
MeSH Terms: conditions — Arthritis, Rheumatoid; Lupus Erythematosus, Systemic

STUDY DESIGN:
Intervention Model Description: Sub-project 1: Randomized crossover study Sub-project 2: Randomized parallel Sub-project 3: Single groupe
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Deep breathing (Experimental): Sub-project 1: To compare the effect of one session of DB and one session of non-invasive auricular tVNS on vagal nerve tone measured by HRV in healthy participants and in patients with RA and SLE.
  Sub-project 2: A dose-response study in healthy participants comparing the effect of 5, 15 and 30 minutes of DB on HRV.
  Sub-project 3: To investigate the effect of the optimal dose found in sub-project 2 in patients with RA and SLE measured by HRV, and to investigate its reproducibility by doing it twice.
  Interventions: Device: Non-invasive auricular electrical transcutaneous vagus nerve stimulation; Other: Deep breathing

INTERVENTIONS:
Device: Non-invasive auricular electrical transcutaneous vagus nerve stimulation — A NEMOS ® stimulator (Cerbomed, Erlangen, Germany) is used for transcutaneous auricular vagus nerve stimulation. This is a handheld battery driven stimulator which stimulates conca in the outer ear. It stimulates in a serie of small electrical impulses with a pulse width at 250 us and a frequency at 25 Hz for 30 minutes in a cycle for 30 seconds "on" and 30 seconds "off" to avoid habituation. It is previously indicated that a stimulation intensity at 0,5 mA, 1 mA or 1,5 mA does not cause a significant chance in HRV, thus 0,5 mA is used in this study.
Other: Deep breathing — The participant is first verbally introduced to the breathing exercises, and then to the visually cue (animation), which the participant have to follow throughout the session.

SUMMARY:
This interventional study aims to investigate the effect of deep breathing (DB) and transcutaneous electrical vagus nerve stimulation (tVNS) on heart rate variability (HRV) in healthy participants and patients with rheumatoid arthritis (RA) or systemic lupus erythematosus (SLE). HRV is used as a surrogate measure of vagal nerve tone.

The study consists of three sub-projects:

Sub-project 1: To compare the effect of one session of DB and one session of non-invasive auricular tVNS on vagal nerve tone measured by HRV in healthy participants and in patients with RA and SLE. The hypotheses is that DB has a similar effect on HRV as non-invasive electrical tVNS.

Sub-project 2: A dose-response study in healthy participants comparing the effect of 5, 15 and 30 minutes of DB on HRV. The hypothesis was that HRV increases as a function of the number of minutes the DB is performed in healthy participants.

Sub-project 3: To investigate the effect of the optimal dose found in sub-project 2 in patients with RA and SLE measured by HRV, and to investigate its reproducibility by doing it twice.The hypothesis was that HRV increases after DB in patients with RA and SLE, and the effect is reproducible.

In all three sub-projects the washout period will be investigated by measuring HRV three times after the intervention. We hypothesise that the effect of DB and tVNS on HRV decreases over time.

ELIGIBILITY:
Inclusion Criteria:

* Men and women in the age range from 18 years to 85 years old.
* For subproject 1 and 3 the participants must be diagnosed with either rheumatoid arthritis or systemic lupus erythematosus.
* Must sign and date informed consent.

Exclusion Criteria:

* Lacking ability to make or understand informed consent.
* Medical history with psychiatric or psychological conditions which the person in charge of the research estimates will affect the participants ability to participate in the study.
* Furthermore participants with severe mental illness will be excluded due to the fact that severe mental illness cause decreased heart rate variability.
* Pregnancy.
* Addict or prior addict defined as abuse of hash, opioids or other euphoriant drugs.
* Known atrial fibrillation or atrial flutter.
* Known chronic lung disease.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2021-09-01 (Actual); Primary Completion 2022-09 (Estimated); Study Completion 2022-09 (Estimated)

PRIMARY OUTCOMES:
Heart rate variability root mean square of successive R-R intervals (RMSSD) | HRV is measured with five ECG recordings, each lasting 5 min. Two measurements with 5 minutes apart are made just prior to the 30 minutes of deep breathing/tvns. Three measurements are made after the intervention, separated by 7,5 minutes each.
  Heart rate variability is used as a surrogate measure of vagus nerve activity. The primary outcome is changes in the HRV-parameter RMSSD

SECONDARY OUTCOMES:
Heart rate variability standard deviation of the R-R intervals (SDNN) and pairs of successive R-R intervals that differ more than 50 milliseconds divided by the total number of R-R intervals (PNN50) | HRV is measured before and after 30 minutes of deep breathing/tvns.
  Heart rate variability is used as a surrogate measure of vagus nerve activity - change in PNN50, SDNN

CONTACTS AND LOCATIONS:
Overall Officials: Salome Kristensen, MD, PhD, Principal Investigator — Aalborg University Hospital
Locations (1):
- Aalborg Universitetshospital, Aalborg, North Denmark, Denmark